CLINICAL TRIAL: NCT02548884
Title: Pancreatic Sphincterotomy Versus Double Wire Technique in Difficult Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Leena Kylanpaa, M.D, Ph.D, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Difficult cannulation
Record Dates: First submitted 2015-09-03; First posted 2015-09-14 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pancreatic sphincterotomy (Active Comparator): Pancreatic sphincterotomy technique used in difficult biliary cannulation
  Interventions: Procedure: Biliary cannulation
- Double guide wire (Active Comparator): Double guide wire technique used in difficult biliary cannulation
  Interventions: Procedure: Biliary cannulation

INTERVENTIONS:
Procedure: Biliary cannulation

SUMMARY:
The purpose of the study is to compare two different techniques (pancreatic sphincterotomy (PS) and double wire technique (DGW)) regarding the risk of post-ERCP pancreatitis (PEP) and the success of cannulation in difficult cannulation. For the study, the difficult cannulation is de-fined as situation when the common bile duct has not been cannulated in five minutes, after five attempts or after two pancreatic guide wire passages or when any of those limits is exceeded. The two techniques, the PS and the DGW, will be compared in random fashion. The primary end-point is the risk of PEP .

ELIGIBILITY:
Inclusion Criteria:

* Naive papilla, ERCP indication common bile duct cannulation

Exclusion Criteria:

* No consent to the study
* Ongoing pancreatitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1190 (Actual)
Dates: Start 2015-09; Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Post ERCP pancreatitis defined by ESGE guidelines published 2014 | 48 hours
  Acute pancreatitis within 48 hours post ERCP. Post-ERCP pancreatitis (PEP) is defined as the presence of abdominal pain attributable to acute pancreatitis, together with a need for an unplanned hospitalization or an extension of a planned hospitalization by at least 2 days, and a serum /plasma amylase at least 3 times above the upper limit of normal at 24 hours after the procedure.

SECONDARY OUTCOMES:
Biliary cannulation success within 15 minutes after randomization | 15 minutes
  After randomization, timing to get the wire in biliary duct. First assessed the number of procedures succeeded in 15 minutes.
Biliary cannulation success, total number | 2 hours
  The total number of successful biliary cannulations after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

REFERENCES:
- [Background] Halttunen J, Meisner S, Aabakken L, Arnelo U, Gronroos J, Hauge T, Kleveland PM, Nordblad Schmidt P, Saarela A, Swahn F, Toth E, Mustonen H, Lohr JM. Difficult cannulation as defined by a prospective study of the Scandinavian Association for Digestive Endoscopy (SADE) in 907 ERCPs. Scand J Gastroenterol. 2014 Jun;49(6):752-8. doi: 10.3109/00365521.2014.894120. Epub 2014 Mar 14. PMID 24628493